CLINICAL TRIAL: NCT05617339
Title: Tailored Digital Treatment for Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGFOUREG-979683
Record Dates: First submitted 2022-10-17; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Migraine With Aura; Migraine Without Aura
Keywords: migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The groups are predetermined based on the tool randomizer.org and blinded to the researcher assigning the participants to groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised internet-based treatment "I am". (Experimental): Need-based internet-based treatment
  Interventions: Behavioral: I am (internet approach to migraine)
- Treatment As Usual (No Intervention): Control group, Treatment in primary care which is medical treatment

INTERVENTIONS:
Behavioral: I am (internet approach to migraine) — I AM has a biopsychosocial perspective. Modules 1-3 and 10 are mandatory and for those who are in need of shorter support and module 1-10 is for those who have more frequent and severe migraines and want a long time of support and treatment. The rationale of the treatment assumes that we do not know why we get migraines and instead focus on becoming as good as possible at managing the migraine attacks. The focus area of the treatments cognitive-behavioral interventions is, among other things, psychoeducation, what migraine is and what happens in the body during migraines and pain, interpretation of symptoms and information processing, training to stop through mindfulness and becoming aware of assumptions that guide behavior during pain management, management of grief, worry, guilt and feelings of shame based on self-compassion, challenging avoidances in a valued direction through ACT interventions and physiotherapist-led cardio training and exercises.
  Other Names: Learn to live with migraine (Lär dig leva med migrän)
  Arms: Personalised internet-based treatment "I am".

SUMMARY:
Background: An individualized internet-based treatment program from a biopsychosocial perspective has been developed within the Västra Götaland region (VGR) with funds from the Innovation Fund. The treatment program is called Learn to live with migraine and goes by the abbreviation I AM (Internet Approach to Migraine). I AM is a complement to the medical treatment and focuses on pain management and learning to live as good a life as possible with the disease migraine. During the spring of 2022, I AM has been tested regarding the feasibility of primary care on 29 research subjects in a pilot RCT (DNR 2020-02359). A weighted preliminary assessment shows moderate effect size on mental health, that the participants accept the intervention, and that I AM with recruitment and care process can be carried out in a primary care context. Purpose: An overall purpose of the study is to evaluate the effect of the addition of the internet-based biopsychosocial treatment I AM compared to usual treatment (TREATMENT as usual - TAU) in primary care regarding frequency and severity of migraine attacks, functional level, mental health, quality of life and employment rate with a randomized controlled trial design (RCT). An additional aim is to evaluate whether it is possible to prevent episodic migraine from developing into chronic migraine among those who have episodic migraine at the start of the study via the supplement treatment program I AM. Expected results: The greatest expected benefit of I AM is to reduce the burden and suffering of migraines for all the people affected. AM is also expected to increase the availability of treatment with a biopsychosocial perspective, have a quality-enhancing effect in terms of method and increase the patient's participation in their treatment. An environmental aspect is that neither patient nor therapist need to travel, accessibility also increases for individuals living in smaller communities who receive equal treatment.

DETAILED DESCRIPTION:
An overall purpose of the study is to evaluate in a randomized controlled trial (RCT) the effect of the addition of the internet-based treatment Internet Approach to Migraine (I AM ) compared to usual treatment (Treatment as usual - TAU) in primary care regarding frequency and severity of migraine attacks, functional level, mental health, quality of life and employment rate. An additional aim is to evaluate whether it is possible to prevent episodic migraine, among those who have episodic migraine at the start of the study, from developing into chronic migraine in primary care via the addition of the I AM treatment program for migraine, compared to TAU.

Question / Hypothesis Impact evaluation - primary outcomes1. What effect does I AM have, in comparison with treatment as usual (TAU) regarding the frequency and severity of migraine as well as functional capacity, mental health and quality of life, in follow-up measurement after termination, at 6 months after the end of treatment, and at 1 year and 2 years of follow-up measurement? The hypothesis is that there is an interaction effect and that the participants in I AM at follow-ups have a significantly lower degree of frequency and severity of migraine, as well as better functional ability, mental health and quality of life.2. Is there a significant difference between how many people have developed chronic migraine (measured by cut off of 15 days a month?) in the I AM and TAU groups, respectively? The hypothesis being tested is that the frequency and severity of migraine attacks is not reduced or further developed by the targeted treatment program I AM in comparison with TAU.

Process Evaluation - Secondary outcomes3. What effect does I AM have in comparison to TAU regarding flexibility and acceptance, selfcompassion, mindfulness, degree of pain sensitivitization and confidence in one's ability to engage in physical training? How does the effect of the intervention stand after 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* 18 years and up
* diagnosed episodic or chronic migraine with or without aura 3 or more migraine days a month.
* Access to computer / tablet or smartphone with Bankid and internet connection.

Exclusion Criteria:

* ongoing malignant disease
* other rarer migraine diseases such as cluster headache, basilar migraine, hemiplegis migraine, vestibular migraine and eye migraine
* ongoing moderate to more severe psychiatric problems such as depression, anxiety disorders, neuropsychiatric conditions, psychotic disorders, substance abuse and personality disorders
* Ongoing psychological/physiotherapeutic treatment
* People who cannot read, speak or understand the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test-6 (HIT-6) | Week 1
  Frequency and severity of migraine attacks.Two questions are added in the present study: How many migraine days per month have you had on average in the last 3 months? Estimated on a scale of 1-10 how painful the headache was. 0= no pain and 10= worst imaginable pain. What percentage have you been employed in the last 3 months?
Headache Impact Test-6 (HIT-6) | post (week 8 or 20)
  Frequency and severity of migraine attacks.Two questions are added in the present study: How many migraine days per month have you had on average in the last 3 months? Estimated on a scale of 1-10 how painful the headache was. 0= no pain and 10= worst imaginable pain. What percentage have you been employed in the last 3 months?
Headache Impact Test-6 (HIT-6) | 6 months follow up
  Frequency and severity of migraine attacks.Two questions are added in the present study: How many migraine days per month have you had on average in the last 3 months? Estimated on a scale of 1-10 how painful the headache was. 0= no pain and 10= worst imaginable pain. What percentage have you been employed in the last 3 months?
Headache Impact Test-6 (HIT-6) | 12 months follow up
  Frequency and severity of migraine attacks.Two questions are added in the present study: How many migraine days per month have you had on average in the last 3 months? Estimated on a scale of 1-10 how painful the headache was. 0= no pain and 10= worst imaginable pain. What percentage have you been employed in the last 3 months?
Headache Impact Test-6 (HIT-6) | 24 months follow up
  Frequency and severity of migraine attacks.Two questions are added in the present study: How many migraine days per month have you had on average in the last 3 months? Estimated on a scale of 1-10 how painful the headache was. 0= no pain and 10= worst imaginable pain. What percentage have you been employed in the last 3 months?

SECONDARY OUTCOMES:
Mental Health Continuum Short Form (MHC-SF). | Week 1
  Mental health and quality of life
Mental Health Continuum Short Form (MHC-SF). | post (week 8 or 20)
  Mental health and quality of life
Mental Health Continuum Short Form (MHC-SF). | 6 months follow up
  Mental health and quality of life
Mental Health Continuum Short Form (MHC-SF). | 12 months follow up
  Mental health and quality of life
Mental Health Continuum Short Form (MHC-SF). | 24 months follow up
  Mental health and quality of life
Swedish version of CORE-10 | Week 1
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Swedish version of CORE-10 | up to week 4 or 10.
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Swedish version of CORE-10 | post (week 8 or 20)
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Swedish version of CORE-10 | 6 months follow up
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Swedish version of CORE-10 | 12 months follow up
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Swedish version of CORE-10 | 24 months follow up
  A broader measure of mental health in terms of well-being, symptoms, function and risk.
Self-Efficacy for Exercise Scale | Week 1
  Their ability to conduct physical exercise
Self-Efficacy for Exercise Scale | up to week 4 or 10.
  Their ability to conduct physical exercise
Self-Efficacy for Exercise Scale | post (week 8 or 20)
  Their ability to conduct physical exercise
Self-Efficacy for Exercise Scale | 6 months follow up
  Their ability to conduct physical exercise
Self-Efficacy for Exercise Scale | 12 months follow up
  Their ability to conduct physical exercise
Self-Efficacy for Exercise Scale | 24 months follow up
  Their ability to conduct physical exercise
Five Facet Mindfulness Questionnaire | Week 1
  Conscious
Five Facet Mindfulness Questionnaire | post (week 8 or 20)
  Conscious
Five Facet Mindfulness Questionnaire | 6 months follow up
  Conscious
Five Facet Mindfulness Questionnaire | 12 months follow up
  Conscious
Five Facet Mindfulness Questionnaire | 24 months follow up
  Conscious
Self-Compassion Scale | Week 1
  Self compassion
Self-Compassion Scale | post (week 8 or 20)
  Self compassion
Self-Compassion Scale | 6 months follow up
  Self compassion
Self-Compassion Scale | 12 months follow up
  Self compassion
Self-Compassion Scale | 24 months follow up
  Self compassion
Two questions to Haskell 2007 - | Week 1
  Physical activity Physical activity
Two questions to Haskell 2007 - | up to week 20
  Physical activity Physical activity
Two questions to Haskell 2007 - | post (week 8 or 20)
  Physical activity Physical activity
Two questions to Haskell 2007 - | 6 months follow up
  Physical activity Physical activity
Two questions to Haskell 2007 - | 12 months follow up
  Physical activity Physical activity
Two questions to Haskell 2007 - | 24 months follow up
  Physical activity Physical activity
Central Sensitization Inventory (CSI) | Week 1
  Key symptoms associated with central sensitization
Central Sensitization Inventory (CSI) | post (week 8 or 20)
  Key symptoms associated with central sensitization
Central Sensitization Inventory (CSI) | 6 months follow up
  Key symptoms associated with central sensitization
Central Sensitization Inventory (CSI) | 12 months follow up
  Key symptoms associated with central sensitization
Central Sensitization Inventory (CSI) | 24 months follow up
  Key symptoms associated with central sensitization
Acceptance of the treatment | Post (week 8 or 20)
  Acceptance of the treatment Measured with its own constructed form developed for the study. The form consists of four questions: Would you recommend the processing to someone else? How meaningful have you experienced the treatment scale 1-7, as well as two open questions answered in writing: what have you got out of the treatment? What has been less good about the treatment?
Acceptance of the treatment | 6 months follow up
  Acceptance of the treatment Measured with its own constructed form developed for the study. The form consists of four questions: Would you recommend the processing to someone else? How meaningful have you experienced the treatment scale 1-7, as well as two open questions answered in writing: what have you got out of the treatment? What has been less good about the treatment?
Acceptance of the treatment | 12 months follow up
  Acceptance of the treatment Measured with its own constructed form developed for the study. The form consists of four questions: Would you recommend the processing to someone else? How meaningful have you experienced the treatment scale 1-7, as well as two open questions answered in writing: what have you got out of the treatment? What has been less good about the treatment?
Acceptance of the treatment | 24 months follow up
  Acceptance of the treatment Measured with its own constructed form developed for the study. The form consists of four questions: Would you recommend the processing to someone else? How meaningful have you experienced the treatment scale 1-7, as well as two open questions answered in writing: what have you got out of the treatment? What has been less good about the treatment?
Other treatment | post (week 8 or 20)
  "Other treatment" is measured with the question: Have you since you finished the treatment I AM, Learn to live with migraine or since the last self-assessment received other treatment for migraine? If yes, please describe which one.
Other treatment | 6 months follow up
  "Other treatment" is measured with the question: Have you since you finished the treatment I AM, Learn to live with migraine or since the last self-assessment received other treatment for migraine? If yes, please describe which one.
Other treatment | 12 months follow up
  "Other treatment" is measured with the question: Have you since you finished the treatment I AM, Learn to live with migraine or since the last self-assessment received other treatment for migraine? If yes, please describe which one.
Other treatment | 24 months follow up
  "Other treatment" is measured with the question: Have you since you finished the treatment I AM, Learn to live with migraine or since the last self-assessment received other treatment for migraine? If yes, please describe which one.
Bulls eye | Week 1
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).
Bulls eye | up to week 20
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).
Bulls eye | post (week 8 or 20)
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).
Bulls eye | 6 months follow up
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).
Bulls eye | 12 months follow up
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).
Bulls eye | 24 months follow up
  Behavioral activation in a valued direction was measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal &melin, 2012). The self-assessment scale is divided into four areas of values in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good kriterieva deaths (Lundgren, Dahl &hayes, 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- FoU primary care Södra Älvsborg, Borås, Sven Eriksonsplatsen 4, Sweden